CLINICAL TRIAL: NCT01075867
Title: Multi-dimensional Prevention Program After Acute Coronary Syndrome (ELIPS) (SPUM-ACS- SP1)
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, François MACH, Pr, University of Bern
Other Study IDs: SPUM-ACS-SP1
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control group: Before ELIPS implementation 12 months follow-up
- Treatment group: After ELIPS implementation 12 months follow-up

SUMMARY:
To demonstrate the effectiveness of the ELIPS programme (Multi-dimEnsionaL preventIon Program after Acute coronary Syndrome), which aims at improving quality of care of patients admitted to hospital with Acute Coronary Syndrome (ACS) in the Swiss setting. The program targets an increase in prescription rates by physicians and long term medication adherence and adoption of healthy lifestyle attitudes by patients.

The program is dedicated to caregivers to increase their application of guidelines into practice, to increase their confidence in therapeutic education of patients, and to patients to improve their understanding of ACS and its treatment and to increase their motivation for long term treatment,.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years
* Admitted for an ACS, that is with symptoms compatible with angina pectoris (chest pain, breathlessness) and at least one of the following 3 features : a) Elevation or depression of the ST segment, inverted T waves or dynamic changes in the repolarization phase b) Positive troponin c) Known coronary artery disease. A significant coronary artery disease must be confirmed angiographically.

Exclusion Criteria:

* Severe physical disability or dement
* Less than 1 year of life expectancy for non cardiac reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Admitted for an Acute Coronary Syndrome
Sampling Method: Probability Sample
Enrollment: 2498 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
composite of death and cardiovascular event | 1 year
  Composite of
  * death from any cause,
  * myocardial infarction,
  * documented unstable angina requiring rehospitalization,
  * revascularization (performed at least 30 days after randomization),
  * documented new or worsen lower limb ischemia,
  * stroke
  * transient cerebral ischemic accident.

SECONDARY OUTCOMES:
Process outcome at discharge | 1 year
  Prescription of recommended treatment at discharge:
  * Cardiovascular medication (Lipid lowering treatment, beta-blockers, antithrombotic therapy (acetylsalicylic acid, clopidogrel), ACE-inhibitors, AT-II antagonists)
  * Smoking cessation counseling during hospital stay
  * Referral to cardiovascular rehabilitation center
  * Use of educational booklet at discharge
Clinical outcomes at follow-up | 1 year
  Individual data on each of the composite outcome
  Cardiovascular mortality
Surrogate outcomes at follow-up | 1 year
  Cardiovascular risk factor control at follow-up:
  * arterial blood pressure,
  * fasting blood glucose,
  * blood lipids (LDL-Cholesterol, HDL-Cholesterol, Triglycerides),
  * smoking cessation (7-days point prevalence at one year and continuous abstinence since hospitalisation)
  * body mass index reduction
  * abdominal waist reduction
  Quality of life and utility (EQ-5D questionnaire) Adherence to medication (MAS questionnaire) Physical activity (IPAQ questionnaire) Motivation to adopt therapeutic lifestyle attitudes (smoking cessation, diet change, physical activity)

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - University Hospital, Bern
  - University Hospitals, Geneva
  - University Hospital, Lausanne
  - University Hospital,, Zurich

REFERENCES:
- [Derived] Weidmann L, Obeid S, Mach F, Shahin M, Yousif N, Denegri A, Muller O, Raber L, Matter CM, Luscher TF. Pre-existing treatment with aspirin or statins influences clinical presentation, infarct size and inflammation in patients with de novo acute coronary syndromes. Int J Cardiol. 2019 Jan 15;275:171-178. doi: 10.1016/j.ijcard.2018.10.050. Epub 2018 Oct 16. PMID 30344063
- See also: Related Info — http://www.spum-acs.ch